CLINICAL TRIAL: NCT03084614
Title: CD8 Reactivity to Microorganisms in Blood and Breast Milk
Status: Terminated | Type: Observational
Why Stopped: Slow/insufficient accrual
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170068; 17-I-0068
Record Dates: First submitted 2017-03-15; First posted 2017-03-21 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Immune Modulation; Tuberculosis; Leprosy; Pertussis; Lyme Disease
Keywords: Infectious Diseases; Dendritic Cells; Pathogens; Passive Cellular Immunity
MeSH Terms: conditions — Tuberculosis; Leprosy; Whooping Cough; Lyme Disease; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Controls: non exposed controls
- donors with naturally enriched antimicrobial blood samples and: Donors with naturally enriched antimicrobial blood samples an breast milk, Comparisons will be made with non exposed controls.

SUMMARY:
Background:

When a person is exposed to something that causes an infection, the body sends a type of cell called CD8 T cells to attack it. Those cells are also found in breast milk. Nursing mothers pass these cells to their child, which helps the child fight infections, too. Researchers want to learn more about how CD8 cells work to keep people healthy.

Objective:

To learn more about how the human body fights off infections.

Eligibility:

People age 18 years and older who either have an infection, are suspected to have an infection, or recently got a vaccine.

The household contacts of these people and people who have not been recently exposed to any infection are also needed.

Design:

Participants will be screened with a medical and health history and physical exam. They may have blood tests.

The first study visit can be the same day as screening. It can be up to 3 months later. For those visits, screening tests will be repeated.

At the first visit, participants will have blood collected from an arm vein.

Participants who are breastfeeding may provide a small sample of breast milk. They may collect it at home or bring a pumping device to NIH to collect it. NIH can also provide a breast pump.

Participants may be contacted for up to 1 year after the first visit to give samples of blood and/or breast milk.

Up to 4 additional visits, which will each take about 1 hour, may be scheduled.

A personal physician or local lab can collect blood from participants and ship it to NIH. Breast milk cannot be shipped.

DETAILED DESCRIPTION:
Cellular lysates from purified protein derivative-positive donors have been reported to transfer tuberculin reactivity to na(SqrRoot) ve recipients, but not diphtheria reactivity; similarly, cell lysates from diphtheria-reactive donors appear to transfer diphtheria reactivity without impacting responses to tuberculin. A historically controversial topic, the terms transfer factor and dialyzed leukocyte extract were used to characterize the reactivity-transferring properties of lysates. We found that the cellular extract derived from antigen-specific memory CD8+ T cells induces interleukin (IL)-6 from antigen-matched antigen-presenting cells. This ultimately elicits IL-17 from bystander memory CD8+ T cells. We identified that dialyzable peptide sequences, S100a9, and the TCR <= chain from CD8+ T cells contribute to the molecular nature of this activity. We further showed that extracts from antigen-targeted T cells enhance immunity to Staphylococcus aureus and Candida albicans. The observed anti-Candida activity of lysates was enhanced when the cells were taken from individuals with higher-than-average exposure to Candida and correlated with increased numbers of Candida-reactive T-cells. These effects are sensitive to immunization protocols and extraction methodology in ways that may explain past discrepancies in the reproducibility of passive cellular immunity. Work by other groups has revealed that memory CD8+ T cells are also the only cell population enriched in breast milk as compared to an equal volume of peripheral blood. Taken together, it may be that the CD8+ memory T cells in breast milk serve as a mechanism of passive cellular immunity transference from mother to offspring. We thus aim to expand our analysis into the potential that lysates taken from sources with enriched immunity against a given microorganism will induce greater in vivo and mouse model activity compared to lysates from non-immune sources, and that this difference in lysate activity will be directly related to the CD8+ T cell enrichment.

In this study, we will collect blood and/or breast milk samples from donors with known or suspected exposure to pathogens, and also from healthy non-exposed volunteers. Research evaluations of samples will be done for the relevant microbe(s) of interest. The volume of blood taken from lacting mothers will be limited to 20mL or less per visit. Cells may be proliferated, immortalized, lysed and dialyzed, and/or stored. Cellular lysates will subsequently be used in both in vitro and pre-clinical animal models to assess for therapeutic potential.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Age 18+ years.
2. Willing to allow storage of blood, breast milk, and cells for future research.
3. Willing to have genetic testing performed.
4. Meets one of the 3 following criteria:

   1. Confirmed exposure:

      -Exposure has been verifiably documented (eg, receiving an immunization or DNCB sensitization treatment).

      OR

      -Clinical history is consistent with established epidemiology of the microbe of interest (eg, documentation of past infection; or to a lesser priority travel to endemic areas or living with an individual that suffers from chronic infection with the targeted microbe).

      AND

      -Positive results on established clinical immunity tests (eg, viral RNA, antibody titers, etc).
   2. Suspected exposure: Clinical history is consistent with established epidemiology of the microbe of interest (eg, travel to endemic areas, documentation of past infection) but no established clinical assay exists to verify exposure.
   3. Non-exposed: Absence of exposure to targeted microorganisms as measured by lack of exposure to infected individuals, lack of travel to endemic areas, no immunization history, negative screening tests, or other methods of establishing exposure history to mucosal microbial agents.

EXCLUSION CRITERIA:

1. Active use of immunosuppressive medications.
2. Any condition that, in the opinion of the investigator, contraindicates participation in this study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: clinical center patients, family members, healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2018-02-16 (Actual); Study Completion 2019-11-08 (Actual)

PRIMARY OUTCOMES:
To compare the in vitro and mouse model immune stimulatoryproperties of lysates derived from microbe-specific CDB+ T cellenriched sources. | There are no definitive time points in this sample collection study

SECONDARY OUTCOMES:
To compare how the in vitro and mouse model immune stimulatoryproperties of breast milk vary with the microbe specific CDB+ T cellconcentration. | There are no definitive time points in this sample collection study

CONTACTS AND LOCATIONS:
Overall Officials: Ian A Myles, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Myles IA, Zhao M, Nardone G, Olano LR, Reckhow JD, Saleem D, Break TJ, Lionakis MS, Myers TG, Gardina PJ, Kirkpatrick CH, Holland SM, Datta SK. CD8+ T cells produce a dialyzable antigen-specific activator of dendritic cells. J Leukoc Biol. 2017 Jan;101(1):307-320. doi: 10.1189/jlb.3A0216-082R. Epub 2016 Aug 11. PMID 27515950
- [Background] Viza D, Fudenberg HH, Palareti A, Ablashi D, De Vinci C, Pizza G. Transfer factor: an overlooked potential for the prevention and treatment of infectious diseases. Folia Biol (Praha). 2013;59(2):53-67. doi: 10.14712/fb2013059020053. PMID 23746171
- [Background] Chahroudi A, Cartwright E, Lee ST, Mavigner M, Carnathan DG, Lawson B, Carnathan PM, Hashempoor T, Murphy MK, Meeker T, Ehnert S, Souder C, Else JG, Cohen J, Collman RG, Vanderford TH, Permar SR, Derdeyn CA, Villinger F, Silvestri G. Target cell availability, rather than breast milk factors, dictates mother-to-infant transmission of SIV in sooty mangabeys and rhesus macaques. PLoS Pathog. 2014 Mar 6;10(3):e1003958. doi: 10.1371/journal.ppat.1003958. eCollection 2014 Mar. PMID 24604066